CLINICAL TRIAL: NCT04872764
Title: The Effect of Acute Kidney Injury on Prognosis in Patients Hospitalised for COVID-19.
Brief Title: Acute Kidney Injury in Patients With CoVID-19
Acronym: AKI-COVID-19
Status: Completed | Type: Observational
Sponsor: Uşak University (Other)
Responsible Party: Principal Investigator, Zelal Adibelli, Asistant Professor, Uşak University
Other Study IDs: UsakU3
Record Dates: First submitted 2021-05-02; First posted 2021-05-04 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Covid19; Acute Kidney Injury
MeSH Terms: conditions — COVID-19; Acute Kidney Injury | interventions — Mortality

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 patients with acute kidney injury: COVID-19 patients with acute kidney injury
  Interventions: Other: duration of hospitalization, mortality rate
- COVID-19 patients without acute kidney injury: COVID-19 patients without acute kidney injury
  Interventions: Other: duration of hospitalization, mortality rate

INTERVENTIONS:
Other: duration of hospitalization, mortality rate — duration of hospitalization, mortality rates of patients hospitalised for COVID-19 evaluated and compared in patients with and without acute kidney injury.

SUMMARY:
We aimed to investigate the effect of Acute Kidney Injury (AKİ) on the prognosis of patients hospitalised for COVID-19.

DETAILED DESCRIPTION:
The effect of Acute Kidney Injury (AKİ) on the prognosis of patients hospitalised for COVID-19. Patients hospitalised for COVID-19 and acute kidney injury will be enrolled. The duration of hospitalisation, mortality rates will be compared in COVID-19 patients with and without acute kidney injury.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalised with COVID-19.
* Patients hospitalised with COVID-19 with Acute Kidney Injury

Exclusion Criteria:

-

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients hospitalised for COVID-19 with and without acute kidney injury
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
mortality rate | 6 months
  mortality rates of COVID-19 patients with and without Acute Kidney Injury
duration of hospitalisation | 6 months
  time between admission to hospital and discharge for COVID-19 patients with and without Acute Kidney Injury

CONTACTS AND LOCATIONS:
Overall Officials: Zelal Adibelli, Principal Investigator — Uşak University
Locations (1):
- Usak University, Uşak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No